CLINICAL TRIAL: NCT02060487
Title: A MULTINATIONAL, MULTICENTER STUDY TO ASSESS THE EFFECTS OF ORAL SILDENAFIL ON MORTALITY IN ADULTS WITH PULMONARY ARTERIAL HYPERTENSION (PAH)
Brief Title: Effects of Oral Sildenafil on Mortality in Adults With PAH
Acronym: AFFILIATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated by Sponsor at recommendation of Data Monitoring Committee after completion of first interim analysis as primary objective was met.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1481324; 2013-004362-34 (EudraCT Number); AFFILIATE (Other: Alias Study Number)
Record Dates: First submitted 2014-01-29; First posted 2014-02-12 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; pulmonary hypertension; PAH; sildenafil; revatio
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: sildenafil citrate
- Medium dose (Experimental)
  Interventions: Drug: sildenafil citrate
- High dose (Experimental)
  Interventions: Drug: sildenafil citrate

INTERVENTIONS:
Drug: sildenafil citrate — sildenafil citrate (PDE-5 inhibitor) 5 mg tablet TID until study treatment discontinued or end of study
  Other Names: Revatio
  Arms: Low dose
Drug: sildenafil citrate — sildenafil citrate (PDE-5 inhibitor) 20 mg tablet TID until study treatment discontinued or end of study
  Other Names: Revatio
  Arms: Medium dose
Drug: sildenafil citrate — sildenafil citrate (PDE-5 inhibitor) 80 mg tablet TID until study treatment discontinued or end of study
  Other Names: Revatio
  Arms: High dose

SUMMARY:
This is a blinded study in adult patients with PAH evaluating the relative effects of sildenafil on mortality when administered at the three doses (80 mg, 20 mg or 5 mg, all three times per day [TID]). In addition, the relative effects on clinical worsening and 6-minute walking distance (6MWD) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects ≥ 18 <75 years of age with any of the following conditions:

* Idiopathic Primary Pulmonary Arterial Hypertension (IPAH)
* PAH secondary to connective tissue disease
* PAH with surgical repair (at least 5 years previously) of atrial septal defect (ASD),ventricular septal defect (VSD), patent ductus arteriosus (PDA) and aorto-pulmonary window
* PAH diagnosis confirmed by right heart catheterization performed within 12 months prior to randomization
* Functional Class II-IV; Baseline 6MWD ≥ 50 m.

Exclusion Criteria:

* Significant (ie, >2+) valvular disease other than tricuspid regurgitation or pulmonary regurgitation
* History of cardiac arrest, respiratory arrest, hemodynamic collapse, CPR, ventricular tachycardia, ventricular fibrillation, or uncontrolled atrial fibrillation
* History of pulmonary embolism; History of chronic lung disease / restrictive lung disease (eg, chronic obstructive pulmonary disease (COPD) or scleroderma) with impairment of lung function
* No prior long term treatment with PDE-5 inhibitors
* Treatment with bosentan OR riociguat within 3 months of randomization
* Current treatment with nitrates or nitric oxide

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-09-22 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (11):
  - Emory University Investigational Drug Services, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Frederik Meijer Heart & Vascular Institute Cardiovascular Research, Grand Rapids, Michigan
  - Spectrum Health Butterworth Hospital IDS Pharmacy, Grand Rapids, Michigan
  - Spectrum Health Heart & Lung Specialized Care Clinic, Grand Rapids, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Spectrum Health Medical Group - Pulmonary Division, Grand Rapids, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Robert V. Sibilia MD, Inc., Wooster, Ohio
  - UT Southwestern Medical School, Dallas, Texas
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (4):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Australian Respiratory and Sleep Medicine Institute, Bedford Park, South Australia
- University Hospital of Mont-Godinne, Yvoir, Belgium
- Bosnia and Herzegovina (4):
  - University Clinical Center of the Republic of Srpska, Banja Luka, B&h/republic of Srpska
  - Clinical Center University Sarajevo, Sarajevo, Bosnia and Herzegovina/canton Sarajevo
  - Health Institution Special Hospital "Medical Institute Bayer", Tuzla, Canton Tuzla
  - University Clinical Hospital Mostar, Mostar, Herzegovina-neretva Canton
- Croatia (2):
  - University Hospital Center Zagreb, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (3):
  - Vseobecna fakultni nemocnice v Praze, Prague, Czech Republic
  - Fakultni nemocnice Olomouc, Olomouc
  - Institut Klinicke a Experimentalni Mediciny, Prague
- Germany (7):
  - DRK Kliniken Berlin, Westend, Berlin
  - Universitaetsklinikum der TU Dresden, Dresden
  - Universitatsklinikum TU Dresden, Dresden
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Thoraxklinik am Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
- Greece (4):
  - University General Hospital of Athens "Attikon", Athens, Attica
  - University General Hospital of Alexandroupolis, Alexandroupoli, Evros
  - University General Hospital of Patras, Pátrai
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Malaysia (4):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Serdang, Kajang, Selangor
  - University Malaya Medical Centre, Kuala Lumpur
- Mexico (3):
  - Centro De Prevencion Y Rehabilitacion De Enfermedades Pulmonares Crónicas, Monterrey, Nuevo León
  - Centro de Desarrollo Biomedico, Mérida, Yucatán
  - Centro de Estudios Clinicos de Queretaro S.C., Querétaro
- Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin, Poland
- Romania (2):
  - Institutul Inimii ,,Niculae Stancioiu" Cluj Napoca, Cluj-Napoca
  - Institutul de Urgenta pentru Boli Cardiovasculare si Transplant Targu-Mures, Târgu Mureş
- Russia (4):
  - FSBI "V.A. Almazov National Medical Research Center", Saint Petersburg, Russian Federation
  - FSBI "Research Institute of complex problems of cardiovascular diseases", Kemerovo
  - FSBI Scientific Research Institute of Pulmonology of FMBA, Moscow
  - FSBI "E.Meshalkin National medical research center", Novosibirsk
- Serbia (5):
  - Institute for Cardiovascular disease of Vojvodina, Kamenitz, Vojvodina
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz, Vojvodina
  - Clinical Center of Serbia, Belgrade
  - University Medical Center Zvezdara, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Singapore (2):
  - National University Heart Centre, National University Hospital Singapore (NUHS), Singapore
  - Khoo Teck Puat Hospital, Singapore
- South Africa (2):
  - Center of Chest Diseases, Johannesburg, Gauteng
  - Dr PG Williams Practice, Johannesburg, Gauteng
- Hospital Universitario Vall d´Hebrón, Barcelona, Catalonia, Spain
- Thailand (7):
  - Faculty of Medicine, Chulalongkorn University, Pathumwan, Bangkok
  - King Chulalongkorn Memorial Hospital, Faculty of Medicine, Chulalongkorn University, Pathumwan, Bangkok
  - Division of Cardiology, Department of Medicine, Faculty of Medicine, Khon Kaen University, Muang District, Changwat Khon Kaen
  - Queen Sirikit Heart Center of the Northeast, Khon Kaen University, Muang District, Changwat Khon Kaen
  - Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Muang District, Changwat Khon Kaen
  - Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai
  - Division of Cardiology, Department of Internal Medicine, Faculty of Medicine, Chiang Mai University, Sripoom Sub-district, Muang, Chiang Mai
- Turkey (Türkiye) (5):
  - Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Bakirkoy
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul, Fatih
  - Istanbul University Haseki Cardiology Institute, Istanbul, Fatih
  - Dokuz Eylul Üniversitesi Tıp Fakültesi Kardiyoloji Bilim Dalı, Izmir, Inciralti
  - Marmara University Pendik Training and Research Hospital, Istanbul, Pendik
- Ukraine (6):
  - Komunalne nekomertsiine pidpryiemstvo, Kharkiv
  - Komunalne nekomertsiine pidpryiemstvo Oleksandrivska klinichna likarnia m. Kyieva, Kyiv
  - Komunalne nekomertsiine pidpryiemstvo, Kyiv
  - Derzhavna ustanova Natsionalnyi naukovyi tsentr, Kyiv
  - Komunalne pidpryiemstvo "Dnipropetrovskyi oblasnyi klinichnyi tsentr kardiolohii ta kardiokhirurhii", M. Dnipro
  - Komunalne nekomertsiine pidpryiemstvo, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hoeper MM, Ewert R, Jansa P, Sirenko Y, Skride A, Balagtas C, Hackley S, Vogt S, Abreu P, Haughie S, Hassan T, Oudiz RJ. Randomized, Multicenter Study to Assess the Effects of Different Doses of Sildenafil on Mortality in Adults With Pulmonary Arterial Hypertension. Circulation. 2024 Jun 18;149(25):1949-1959. doi: 10.1161/CIRCULATIONAHA.123.068107. Epub 2024 May 16. PMID 38752352
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481324&StudyName=Effects%20of%20Oral%20Sildenafil%20on%20Mortality%20in%20Adults%20with%20PAH

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, parallel-group, multinational and multicenter study to assess the effects of oral sildenafil on mortality in adult participants with pulmonary arterial hypertension (PAH). The study was conducted at 68 active sites in 23 countries.
Groups:
- Sildenafil 5 mg: Participants received a single tablet of sildenafil at a dose of 5 milligram (mg) along with two tablets of placebo matching 20 mg and 80 mg sildenafil orally thrice daily (TID) until discontinuation of study treatment or end of study. The maximum duration of study treatment was 2080 days approximately. Participants were followed up for at least 28 days after last dose of study treatment.
- Sildenafil 20 mg: Participants received a single tablet of sildenafil at a dose of 20 mg along with two tablets of placebo matching 5 mg and 80 mg sildenafil orally TID until discontinuation of study treatment or end of study. The maximum duration of study treatment was 1984 days approximately. Participants were followed up for at least 28 days after last dose of study treatment.
- Sildenafil 80 mg: Participants received a single tablet of sildenafil at a dose of 20 mg along with two tablets of placebo matching 5 mg and 80 mg sildenafil orally TID on day 1 for 2 weeks and then titrated up to 80 mg at week 2 along with two tablets of placebo matching 5 mg and 20 mg sildenafil orally TID until discontinuation of study treatment or end of study. The maximum duration of study treatment was 2073 days approximately. Participants were followed up for at least 28 days after last dose of study treatment.
Period: Overall Study
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg
Started | 129 | 128 | 128
Completed | 0 | 0 | 0
Not Completed | 129 | 128 | 128
Not completed — Other | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 10 | 4
Not completed — Study Terminated By Sponsor | 87 | 89 | 100
Not completed — Randomized in error | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Death | 34 | 25 | 19
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants were included in the baseline analysis population.
Groups:
- Sildenafil 5 mg: Participants received a single tablet of sildenafil at a dose of 5 mg along with two tablets of placebo matching 20 mg and 80 mg sildenafil orally TID until discontinuation of study treatment or end of study. The maximum duration of study treatment was 2080 days approximately. Participants were followed up for at least 28 days after last dose of study treatment.
- Total: Total of all reporting groups
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg | Total
Number analyzed (Participants) | 129 | 128 | 128 | 385
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (15.02) | 51.2 (15.81) | 52.1 (14.72) | 51.6 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 102 | 98 | 297
  Male | 32 | 26 | 30 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 3 | 12
  Not Hispanic or Latino | 124 | 124 | 125 | 373
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 23 | 14 | 19 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 104 | 113 | 108 | 325
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: In this outcome measure number of deaths during the study were reported.
Time Frame: Day 1 of study treatment up to date of death (within a maximum duration of 2102 days)
Population: The intent-to-treat population (ITT) included all randomized participants treated with study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg
Number analyzed (Participants) | 129 | 128 | 128
Participants | 34 | 25 | 19
Statistical Analysis 1: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; Test type: Non-Inferiority — Non-inferiority of sildenafil 20 mg TID versus sildenafil 5 mg TID was to be concluded if the upper limit of the 99.7% confidence interval (CI) for hazard ratio (HR) was less than 2; Hazard Ratio (HR) = 0.68, 99.7% CI 2-sided [0.31 to 1.49] — Hazard ratio estimated from the Proportional Hazards model, stratified by actual previous PAH treatment and etiology of PAH
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 80 mg; Test type: Non-Inferiority — Non-inferiority of sildenafil 80 mg TID vs. sildenafil 5 mg TID was to be concluded if the upper limit of the 99.7% CI for HR was less than 2; Hazard Ratio (HR) = 0.51, 99.7% CI 2-sided [0.22 to 1.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sildenafil 20 mg vs Sildenafil 80 mg; Test type: Non-Inferiority — Non-inferiority of sildenafil 80 mg TID vs. sildenafil 20 mg TID was to be concluded if the upper limit of the 99.7% CI for HR is less than 2; Hazard Ratio (HR) = 0.74, 99.7% CI 2-sided [0.30 to 1.84] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Clinical Worsening Events
Description: Clinical worsening was defined as all-cause mortality, non-elective hospital stay for worsening pulmonary arterial hypertension (PAH) (including but not limited to right heart failure [RHF], initiation of intravenous (IV) prostanoids, lung transplantation, or septostomy) or disease progression. Disease progression was defined as a reduction from baseline in the 6-Minute Walk Distance (6MWD) test by 15% and worsening functional class from baseline, both confirmed by second test within 2 weeks of study treatment.
Time Frame: Day 1 of study treatment up to date of clinical worsening event (within a maximum duration of 2080 days)
Population: ITT population included all randomized participants treated with study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg
Number analyzed (Participants) | 129 | 128 | 128
Participants | 52 | 36 | 28
Statistical Analysis 1: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; Test type: Superiority; p = 0.035, Wald test; Hazard Ratio (HR) = 0.63, 99.7% CI 2-sided [0.33 to 1.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 80 mg; Test type: Superiority; p < 0.001, Wald test; Hazard Ratio (HR) = 0.44, 99.7% CI 2-sided [0.22 to 0.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sildenafil 20 mg vs Sildenafil 80 mg; Test type: Superiority; p = 0.195, Wald test; Hazard Ratio (HR) = 0.72, 99.7% CI 2-sided [0.34 to 1.52] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Month 6
Description: 6MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed. Analysis was performed using mixed model for repeated measures (MMRM), adjusted for baseline 6MWD and for randomization stratification factors: PAH treatment at study entry and etiology of PAH.
Time Frame: Baseline, Month 6
Population: ITT population included all randomized participants treated with study treatment. Here, "overall number of participants analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg
Number analyzed (Participants) | 113 | 118 | 116
Meters | 12.2 [-0.67 to 25.16] | 27.3 [14.52 to 39.99] | 31.2 [18.68 to 43.66]
Statistical Analysis 1: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; Test type: Superiority; p = 0.0627, MMRM; Least-squares means difference = 15.0, 95% CI 2-sided [-0.80 to 30.81]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 80 mg; Test type: Superiority; p = 0.0201, MMRM; Least-squares means difference = 18.9, 95% CI 2-sided [2.99 to 34.86]
Statistical Analysis 3: Comparison: Sildenafil 20 mg vs Sildenafil 80 mg; Test type: Superiority; p = 0.6254, MMRM; Least-squares means difference = 3.9, 95% CI 2-sided [-11.85 to 19.68]

4. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD) at Month 12
Description: as for outcome 3
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Meters
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg
Number analyzed (Participants) | 88 | 89 | 89
Meters | 14.3 [-0.58 to 29.27] | 35.7 [20.91 to 50.48] | 34.8 [20.21 to 49.43]
Statistical Analysis 1: Comparison: Sildenafil 5 mg vs Sildenafil 20 mg; Test type: Superiority; p = 0.0286, MMRM; Least-squares means difference = 21.3, 95% CI 2-sided [2.25 to 40.45]
Statistical Analysis 2: Comparison: Sildenafil 5 mg vs Sildenafil 80 mg; Test type: Superiority; p = 0.0364, MMRM; Least-squares means difference = 20.5, 95% CI 2-sided [1.30 to 39.65]
Statistical Analysis 3: Comparison: Sildenafil 20 mg vs Sildenafil 80 mg; Test type: Superiority; p = 0.9283, MMRM; Least-squares means difference = -0.9, 95% CI 2-sided [-19.94 to 18.19]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study treatment (up to a maximum duration of 2108 days for sildenafil 5 mg; up to a maximum duration of 2012 days for sildenafil 20 mg; up to a maximum duration of 2101 days for sildenafil 80 mg)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. Safety population comprised of all randomized participants treated with study treatment.
Arm/Group | Sildenafil 5 mg | Sildenafil 20 mg | Sildenafil 80 mg
All-Cause Mortality (participants affected / at risk) | 34/129 | 25/128 | 19/128
Serious Adverse Events (participants affected / at risk) | 66/129 | 49/128 | 51/128
Other Adverse Events (participants affected / at risk) | 108/129 | 107/128 | 111/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 5 mg (N=129) | Sildenafil 20 mg (N=128) | Sildenafil 80 mg (N=128)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 3 | 0
Cardiac failure (Cardiac disorders) | 9 | 8 | 3
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 2 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 11 | 4 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 1
Condition aggravated (General disorders) | 1 | 0 | 0
Death (General disorders) | 2 | 0 | 1
Disease progression (General disorders) | 1 | 2 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 3 | 0 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 3
Cellulitis (Infections and infestations) | 2 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0
Leptospirosis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 2
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 6 | 3
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 2 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haemodynamic test (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pleomorphic malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Systemic sclerosis pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug therapy (Surgical and medical procedures) | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 1
Lung transplant (Surgical and medical procedures) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0 | 2
Shock (Vascular disorders) | 1 | 0 | 0
Varicose ulceration (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 5 mg (N=129) | Sildenafil 20 mg (N=128) | Sildenafil 80 mg (N=128)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 11
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypothrombinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 4 | 2
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 2
Atrial flutter (Cardiac disorders) | 3 | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 5 | 5 | 6
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Right ventricular failure (Cardiac disorders) | 3 | 2 | 0
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 5
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 2 | 1
Thyroid malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 3 | 1
Hypoacusis (Ear and labyrinth disorders) | 3 | 1 | 0
Mixed deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 4 | 2
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 4 | 2
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Primary hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0
Asthenopia (Eye disorders) | 1 | 1 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 4 | 0 | 2
Chalazion (Eye disorders) | 0 | 0 | 1
Chromatopsia (Eye disorders) | 0 | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1
Cornea verticillata (Eye disorders) | 0 | 0 | 1
Corneal oedema (Eye disorders) | 1 | 0 | 0
Corneal opacity (Eye disorders) | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0
Dark circles under eyes (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 1 | 1
Dyschromatopsia (Eye disorders) | 0 | 0 | 1
Eye disorder (Eye disorders) | 1 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 2 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 3
Eye pruritus (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 2
Hypermetropia (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 1
Periorbital pain (Eye disorders) | 0 | 0 | 1
Periorbital swelling (Eye disorders) | 0 | 2 | 1
Photophobia (Eye disorders) | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 2
Retinal vascular disorder (Eye disorders) | 0 | 2 | 1
Swelling of eyelid (Eye disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 3 | 2 | 2
Visual impairment (Eye disorders) | 1 | 2 | 4
Visual snow syndrome (Eye disorders) | 0 | 1 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7 | 11
Abdominal symptom (Gastrointestinal disorders) | 1 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 2 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 1 | 1
Dental necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 17 | 20
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 3
Duodenal bulb deformity (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Duodenal vascular ectasia (Gastrointestinal disorders) | 0 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 6 | 10 | 10
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 1 | 3
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 3 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 3 | 2 | 3
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 12 | 8
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 2
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Tongue erythema (Gastrointestinal disorders) | 0 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 5 | 5 | 3
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 10 | 7
Asthenia (General disorders) | 3 | 7 | 2
Catheter site erythema (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 3 | 3 | 0
Chest pain (General disorders) | 7 | 15 | 13
Chills (General disorders) | 2 | 1 | 5
Crying (General disorders) | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 3 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 11 | 10 | 9
Feeling cold (General disorders) | 2 | 1 | 0
Feeling hot (General disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 1 | 0
Ill-defined disorder (General disorders) | 0 | 2 | 0
Inflammation (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 1 | 0
Injection site hypersensitivity (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 2 | 1
Mucosal dryness (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 3 | 2 | 3
Oedema peripheral (General disorders) | 14 | 17 | 8
Pain (General disorders) | 2 | 1 | 3
Peripheral swelling (General disorders) | 7 | 6 | 5
Pyrexia (General disorders) | 3 | 9 | 9
Swelling (General disorders) | 2 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0
Ulcer (General disorders) | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystocholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 2 | 1
Congestive hepatopathy (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 4 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2
Food allergy (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 2 | 1
Multiple allergies (Immune system disorders) | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Secondary immunodeficiency (Immune system disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 3
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bacterial rhinitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 11 | 11 | 8
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 2 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Chronic tonsillitis 0 0 (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 5 | 1 | 6
Cystitis (Infections and infestations) | 3 | 2 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 4 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 1 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 1 | 0
Genital infection female (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 2 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 1 | 2
Herpes virus infection (Infections and infestations) | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0
Incision site abscess (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 6 | 8 | 11
Joint abscess (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 2
Localised infection (Infections and infestations) | 0 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 19 | 16 | 19
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 2
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 3
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 3 | 5
Pulpitis dental (Infections and infestations) | 1 | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 4 | 6
Respiratory tract infection viral (Infections and infestations) | 4 | 5 | 8
Rhinitis (Infections and infestations) | 5 | 5 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 3 | 10
Skin infection (Infections and infestations) | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tongue fungal infection (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 3 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 16 | 8 | 13
Urinary tract infection (Infections and infestations) | 4 | 1 | 5
Vaginal infection (Infections and infestations) | 1 | 1 | 0
Varicella (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 4 | 5 | 3
Viral rhinitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burn oral cavity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Exposure via breast milk (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 3
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Nasal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oral contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood albumin abnormal (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 3 | 3 | 3
Blood cholesterol increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 1
Blood glucose decreased (Investigations) | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 1 | 0
Blood potassium abnormal (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 2
Blood pressure diastolic decreased (Investigations) | 2 | 1 | 1
Blood pressure increased (Investigations) | 3 | 1 | 2
Blood pressure measurement (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 2 | 2
Body temperature increased (Investigations) | 0 | 2 | 1
Breath sounds abnormal (Investigations) | 1 | 0 | 0
Colonoscopy (Investigations) | 1 | 0 | 0
Endoscopy (Investigations) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 1 | 0 | 0
Haemodynamic test (Investigations) | 0 | 2 | 0
Heart rate (Investigations) | 0 | 1 | 0
Heart rate decreased (Investigations) | 1 | 0 | 1
Heart rate increased (Investigations) | 1 | 1 | 0
Heart sounds abnormal (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Protein total abnormal (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1
Staphylococcus test positive (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Ultrasound scan (Investigations) | 0 | 0 | 1
Venous pressure jugular increased (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1
Walking distance test abnormal (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 4 | 1 | 2
Weight increased (Investigations) | 2 | 1 | 1
White blood cell count increased (Investigations) | 0 | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Calcium deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 2 | 1 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 6 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 3 | 2
Mineral metabolism disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 13 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 10 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 10 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 14 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sclerodactylia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Ageusia (Nervous system disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 12 | 15 | 18
Dizziness exertional (Nervous system disorders) | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 26 | 45 | 33
Hypoaesthesia (Nervous system disorders) | 2 | 3 | 2
Hypotonia (Nervous system disorders) | 0 | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Neuritis (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 3 | 2
Postictal paralysis (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 4 | 1
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 3 | 5 | 0
Syncope (Nervous system disorders) | 4 | 4 | 4
Tension headache (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 3
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0
Trigeminal neuritis (Nervous system disorders) | 0 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 0 | 1
Device fastener issue (Product Issues) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 1
Apathy (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 3 | 1
Emotional disorder (Psychiatric disorders) | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 5 | 2
Mental disorder (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 2 | 1 | 3
Renal failure (Renal and urinary disorders) | 1 | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Breast inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 13 | 13
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cancer surgery (Surgical and medical procedures) | 0 | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 1 | 3
Dental operation (Surgical and medical procedures) | 1 | 0 | 0
Haematoma evacuation (Surgical and medical procedures) | 1 | 0 | 0
Myomectomy (Surgical and medical procedures) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 1
Tooth repair (Surgical and medical procedures) | 1 | 0 | 0
Vascular operation (Surgical and medical procedures) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 2
Cyanosis (Vascular disorders) | 1 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 6 | 3 | 4
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 3 | 2
Hyperaemia (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 6 | 5
Hypertensive crisis (Vascular disorders) | 3 | 0 | 0
Hypotension (Vascular disorders) | 9 | 6 | 7
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Labile blood pressure (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Neovascularisation (Vascular disorders) | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 2 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 1
Vasodilatation (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated by Sponsor at recommendation of Data Monitoring Committee after completion of first interim analysis as primary objective was met. For OS and clinical worsening(CW) endpoints, significance level was adjusted to allow for interim analysis. Hence 99.7% CIs were presented instead of 95% CIs. 80mg vs 5mg comparison for OS was primary and it was key secondary for CW. CIs for other dose comparisons for these endpoints were nominal. P-values and CIs for other endpoints were nominal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT02060487/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT02060487/SAP_001.pdf